CLINICAL TRIAL: NCT03722784
Title: Evaluation of the CooperVision, Inc. Invigor A and Invigor B Silicone Hydrogel Daily Wear Contact Lenses When Used for Frequent Replacement for Up to One (1) Month of Daily Wear
Brief Title: Evaluation of Silicone Hydrogel Daily Wear Contact Lenses for Up to One (1) Month of Daily Wear
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: CooperVision, Inc. (Industry)
Responsible Party: Sponsor
Organization: CooperVision International Limited (CVIL) (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: FC160322
Record Dates: First submitted 2018-10-25; First posted 2018-10-29 (Actual); Results first posted 2020-10-01 (Actual); Last update posted 2020-10-01 (Actual); Status verified 2020-08

CONDITIONS: Myopia; Hyperopia; Astigmatism
MeSH Terms: conditions — Myopia; Hyperopia; Astigmatism

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: The subject will know the name of the lens however they will not be aware of which lens is investigational and which lens has been previously cleared. The licensed investigator has not been informed which lens is the investigational lens.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: Yes

ARMS (2):
- Invigor A (test) (Experimental): Subjects will be randomized to wear Invigor A (test) for one month of daily wear during the study.
  Interventions: Device: Invigor A (test)
- Invigor B (Control) (Active Comparator): Subjects will be randomized to wear Invigor B (Control) for one month of daily wear during the study.
  Interventions: Device: Invigor B (control)

INTERVENTIONS:
Device: Invigor A (test) — silicone hydrogel lens
  Arms: Invigor A (test)
Device: Invigor B (control) — silicone hydrogel lens
  Arms: Invigor B (Control)

SUMMARY:
The aim of the study is to evaluate if the performance of Invigor A is substantially equivalent to Invigor B contact lenses when used in a one month recommended replacement, daily wear modality.

DETAILED DESCRIPTION:
This study is a multi-centered, daily wear, monthly replacement, bilateral, randomized in a ratio of two to one (2:1) Test to Control, lens blocked (subjects remain in the same lens brand throughout the study), licensed investigator and subject masked, concurrent controlled study with a study duration of approximately three months evaluating performance equivalence of Invigor A (test) over Invigor B (control) contact lenses.

ELIGIBILITY:
* Inclusion Criteria:

  1. Be at least 18 years of age as of the date of evaluation for the study
  2. Have

     1. Read the informed consent document
     2. Been given an explanation of the informed consent document
     3. indicated understanding of the informed consent document
     4. Signed the informed consent document
  3. Be willing and able to adhere to the instructions provided by the investigational site and be willing to keep all specified appointments.
  4. Be an adapted, frequent replacement, current full - time silicone hydrogel or soft contact lens wearer. An adapted full- time wearer is defined as wearing contact lenses at least 5 days per week for at least 8 hours per day for at least one month prior to participation in the study.
  5. Possess or obtain prior to dispensing, wearable and visually functional (20/40 or better) eyeglasses.
  6. Be in good general health, based on his/her knowledge.
* Exclusion Criteria:

  1. Wearing lenses in a monovision modality and is unwilling to be fit with distance lenses in both eyes for the duration of the study. Note: Subjects may not wear lenses in a monovision modality at any time during the study as it will interfere with the visual acuity analysis.
  2. Poor personal hygiene.
  3. Any active participation in another clinical trial during this trial or within 30 days prior to this study.
  4. To the best of the subject's knowledge, she is currently pregnant, is lactating or is planning a pregnancy within the next 3 months.
  5. A member, relative or household member of the investigator(s) or of the investigational office staff.
  6. A known sensitivity to the ingredients used in the multi-purpose solution approved for use in the study and is unable or unwilling to use the alternate care system.
  7. Had previous refractive surgery; or current or previous orthokeratology treatment.
  8. Aphakic or pseudophakic.
  9. Ocular or systemic disease such as, but not limited to: anterior uveitis or iritis (past or present), glaucoma, Sjögren's syndrome, lupus erythematosus, scleroderma, keratoconus or uncontrolled diabetes.
  10. The need for topical ocular medications or any systemic medication which might interfere with contact lens wear or require the lenses to be removed during the day.
  11. A known history of corneal hypoesthesia (reduced corneal sensitivity), corneal ulcer, corneal infiltrates, iritis, bacterial or fungal infections.
  12. A history of papillary conjunctivitis that has interfered with contact lens wear.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 88 (Actual)
Dates: Start 2018-10-10 (Actual); Primary Completion 2019-01-18 (Actual); Study Completion 2019-06-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Quinn, O.D, Principal Investigator — Quinn, Foster & Associates, OH; Peter Van Hoven, O.D, Principal Investigator — Primary Eyecare group, P.C, TN; Mark Nakano, O.D, Principal Investigator — Mark Nakano, O.D, CA; David Ziegler, O.D, Principal Investigator — Ziegler Leffingwell Eye Center, WI; Cheryl Vincent Riemer, O.D, Principal Investigator — Vision Care Associates, MI; Carmen Castellano, O.D, Principal Investigator — The Koetting Associates, MO
Locations (6):
- United States (6):
  - Mark Nakano. O.D, Torrance, California
  - Vision Care Associates, East Lansing, Michigan
  - The Koetting Associates, St Louis, Missouri
  - Quinn, Foster & Associates, Athens, Ohio
  - Primary Eyecare Group, P.C, Brentwood, Tennessee
  - Ziegler Leffingwell Eye Center, West Allis, Wisconsin

RESULTS

PARTICIPANT FLOW:
Units Other Than Participants: Eyes
Groups:
- Invigor A (Test): Subjects will be randomized in a ratio of two to one (2:1) Test to Control, to wear Invigor A (test) for one month of daily wear during the study.
  Invigor A (test): silicone hydrogel lens
- Invigor B (Control): Subjects will be randomized in a ratio of two to one (2:1) Test to Control, to wear Invigor B (Control) for one month of daily wear during the study.
  Invigor B (control): silicone hydrogel lens
Period: Overall Study
Arm/Group | Invigor A (Test) | Invigor B (Control)
Started | 58; 116 Eyes | 30; 60 Eyes
Completed | 56; 112 Eyes | 28; 56 Eyes
Not Completed | 2; 4 Eyes | 2; 4 Eyes
Not completed — Withdrawal by Subject | 1 | 0
Not completed — Physician Decision | 1 | 1
Not completed — Protocol Violation | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Invigor A (Test): Subjects will be randomized in a ratio of two to one (2:1) Test to Control to wear Invigor A (test) and Invigor B (control) for one month of daily wear during the study.
  Invigor A (test): silicone hydrogel lens
- Invigor B (Control): Subjects will be randomized in a ratio of two to one (2:1) Test to Control to wear Invigor A (test) and Invigor B (control) for one month of daily wear during the study.
  Invigor B (Control): silicone hydrogel lens
- Total: Total of all reporting groups
Arm/Group | Invigor A (Test) | Invigor B (Control) | Total
Number analyzed (Participants) | 58 | 30 | 88
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 58 | 30 | 88
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 33.19 (8.080) | 33.73 (8.497) | 33.38 (8.179)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 39 | 17 | 56
  Male | 19 | 13 | 32
Race/Ethnicity, Customized [Number; unit: participants]
  Black | 2 | 2 | 4
  Chinese | 1 | 0 | 1
  Hispanic/Latino | 4 | 0 | 4
  Japanese | 5 | 3 | 8
  White | 43 | 23 | 66
  Other | 0 | 2 | 2
  Chinese/Japanese | 1 | 0 | 1
  Japanese/Other | 2 | 0 | 2
Region of Enrollment [Number; unit: participants]
  United States | 58 | 30 | 88

OUTCOME MEASURES:

1. Primary Outcome: Number of Eyes With Epithelial Edema - Slit Lamp Findings
Description: Epithelial edema on slit lamp grading scale 0 - 4 (0- No microcysts; normal transparency, 1 Trace - 1 to 20 microcysts; barely discernible local epithelial haziness, 2 Mild - 21 to 50 microcysts; faint but definite localized or generalized haziness, 3 Moderate - 51 to 100 microcysts; significant localized or generalized haziness, 4 Severe - >100 microcysts; definite widespread epithelial cloudiness giving a dull glass appearance to the cornea, or numerous coalescing bullae)
Time Frame: Baseline
Measure: Number; unit: Eyes
Units Other Than Participants: Eyes
Groups:
- Invigor A (Test): Subjects will be randomized in a ratio of two to one (2:1) Test to Control to wear Invigor A (test) for one month of daily wear during the study.
  Invigor A (test): silicone hydrogel lens
- Invigor B (Control): Subjects will be randomized in a ratio of two to one (2:1) Test to Control to wear Invigor B (Control) for one month of daily wear during the study.
  Invigor B (control): silicone hydrogel lens
Arm/Group | Invigor A (Test) | Invigor B (Control)
Number analyzed (Participants) | 56 | 28
Number analyzed (Eyes) | 112 | 56
Eyes
  Grade 0 | 112 | 56
  Grade 1 | 0 | 0
  Grade 2 | 0 | 0
  Grade 3 | 0 | 0
  Grade 4 | 0 | 0

2. Primary Outcome: Number of Eyes With Epithelial Edema - Slit Lamp Findings
Description: as for outcome 1
Time Frame: One Month
Population: Two eyes data was not collected for both test and control lens at the one month visit due to lens discomfort.
Measure: Number; unit: Eyes
Units Other Than Participants: Eyes
Arm/Group | Invigor A (Test) | Invigor B (Control)
Number analyzed (Participants) | 55 | 27
Number analyzed (Eyes) | 110 | 54
Eyes
  Grade 0 | 110 | 54
  Grade 1 | 0 | 0
  Grade 2 | 0 | 0
  Grade 3 | 0 | 0
  Grade 4 | 0 | 0

3. Primary Outcome: Number of Eyes With Stromal Edema - Slit Lamp Findings
Description: Stromal edema on slit lamp grading scale 0-4 (0 None - No edema, 1 Trace - Just detectable clouding, 2 Mild - faint corneal striae, 3 Moderate - Pronounced corneal striae, 4 severe - folds in Descemet's membrane and ≥4 pronounced striae
Time Frame: Baseline
Measure: Number; unit: Eyes
Units Other Than Participants: Eyes
Arm/Group | Invigor A (Test) | Invigor B (Control)
Number analyzed (Participants) | 56 | 28
Number analyzed (Eyes) | 112 | 56
Eyes
  Grade 0 | 112 | 56
  Grade 1 | 0 | 0
  Grade 2 | 0 | 0
  Grade 3 | 0 | 0
  Grade 4 | 0 | 0

4. Primary Outcome: Number of Eyes With Stromal Edema - Slit Lamp Findings
Description: as for outcome 3
Time Frame: One Month
Population: Two eyes data was not collected for both test and control lens at the one month visit due to lens discomfort.
Measure: Number; unit: Eyes
Units Other Than Participants: Eyes
Arm/Group | Invigor A (Test) | Invigor B (Control)
Number analyzed (Participants) | 55 | 27
Number analyzed (Eyes) | 110 | 54
Eyes
  Grade 0 | 110 | 54
  Grade 1 | 0 | 0
  Grade 2 | 0 | 0
  Grade 3 | 0 | 0
  Grade 4 | 0 | 0

5. Primary Outcome: Number of Eyes With Corneal Vascularization - Slit Lamp Findings
Description: Corneal Vascularization on slit lamp grading scale 0-4 (0 None: No vessel penetration, 1 Trace: <1.00 mm vessel penetration, 2 Mild: >1.00 mm to <1.50 mm vessel penetration, 3 Moderate: >1.50 mm to <2.00 mm vessel penetration, 4 Severe: Vessel penetration >2.00 mm) Depth: a. - Epithelial b. - Anterior Stromal c. - Mid/Posterior Stromal Location: N - Nasal T - Temporal I - Inferior S - Superior
Time Frame: Baseline
Measure: Number; unit: Eyes
Units Other Than Participants: Eyes
Arm/Group | Invigor A (Test) | Invigor B (Control)
Number analyzed (Participants) | 56 | 28
Number analyzed (Eyes) | 112 | 56
Eyes
  Grade 0 | 98 | 56
  Grade 1 | 14 | 0
  Grade 2 | 0 | 0
  Grade 3 | 0 | 0
  Grade 4 | 0 | 0

6. Primary Outcome: Number of Eyes With Corneal Vascularization - Slit Lamp Findings
Description: as for outcome 5
Time Frame: One Month
Population: Two eyes data was not collected for both test and control lens at the one month visit due to lens discomfort.
Measure: Number; unit: Eyes
Units Other Than Participants: Eyes
Arm/Group | Invigor A (Test) | Invigor B (Control)
Number analyzed (Participants) | 55 | 27
Number analyzed (Eyes) | 110 | 54
Eyes
  Grade 0 | 98 | 54
  Grade 1 | 12 | 0
  Grade 2 | 0 | 0
  Grade 3 | 0 | 0
  Grade 4 | 0 | 0

7. Primary Outcome: Number of Eyes With Corneal Staining - Slit Lamp Findings
Description: Corneal Staining with fluorescent on slit lamp findings - Present / Absent
Time Frame: Baseline
Measure: Number; unit: Eyes
Units Other Than Participants: Eyes
Arm/Group | Invigor A (Test) | Invigor B (Control)
Number analyzed (Participants) | 56 | 28
Number analyzed (Eyes) | 112 | 56
Eyes
  Present | 10 | 7
  Absent | 102 | 49

8. Primary Outcome: Number of Eyes With Corneal Staining - Slit Lamp Findings
Description: Corneal Staining with fluorescent on slit lamp findings - Present / Absent
Time Frame: One Month
Population: Two eyes data was not collected for both test and control lens at the one month visit due to lens discomfort.
Measure: Number; unit: Eyes
Units Other Than Participants: Eyes
Arm/Group | Invigor A (Test) | Invigor B (Control)
Number analyzed (Participants) | 55 | 27
Number analyzed (Eyes) | 110 | 54
Eyes
  Present | 20 | 9
  Absent | 90 | 45

9. Primary Outcome: Number of Eyes With Corneal Infiltrates - Slit Lamp Findings
Description: Corneal Infiltrates on slit lamp findings - Present / Absent
Time Frame: Baseline
Measure: Number; unit: Eyes
Units Other Than Participants: Eyes
Arm/Group | Invigor A (Test) | Invigor B (Control)
Number analyzed (Participants) | 56 | 28
Number analyzed (Eyes) | 112 | 56
Eyes
  Present | 0 | 0
  Absent | 112 | 56

10. Primary Outcome: Number of Eyes With Corneal Infiltrates - Slit Lamp Findings
Description: Number of Eyes With Corneal Infiltrates on slit lamp findings - Present / Absent
Time Frame: One Month
Population: Two eyes data was not collected for both test and control lens at the one month visit due to lens discomfort.
Measure: Number; unit: Eyes
Units Other Than Participants: Eyes
Arm/Group | Invigor A (Test) | Invigor B (Control)
Number analyzed (Participants) | 55 | 27
Number analyzed (Eyes) | 110 | 54
Eyes
  Present | 0 | 0
  Absent | 110 | 54

11. Primary Outcome: Number of Eyes With Limbal Hyperemia - Slit Lamp Findings
Description: Limbal Hyperemia on slit lamp grading scale 0-4 (0 None: No hyperemia, 1 Trace: Slight limbal hyperemia (mild segmented), 2 Mild: Mild limbal hyperemia (mild circumcorneal), 3 Moderate: Significant limbal hyperemia (marked segmented), 4 Severe: Severe limbal hyperemia (marked circumcorneal).
Time Frame: Baseline
Measure: Number; unit: Eyes
Units Other Than Participants: Eyes
Arm/Group | Invigor A (Test) | Invigor B (Control)
Number analyzed (Participants) | 56 | 28
Number analyzed (Eyes) | 112 | 56
Eyes
  Grade 0 | 112 | 54
  Grade 1 | 0 | 2
  Grade 2 | 0 | 0
  Grade 3 | 0 | 0
  Grade 4 | 0 | 0

12. Primary Outcome: Number of Eyes With Limbal Hyperemia - Slit Lamp Findings
Description: as for outcome 11
Time Frame: One Month
Population: Two eyes data was not collected for both test and control lens at the one month visit due to lens discomfort.
Measure: Number; unit: Eyes
Units Other Than Participants: Eyes
Arm/Group | Invigor A (Test) | Invigor B (Control)
Number analyzed (Participants) | 55 | 27
Number analyzed (Eyes) | 110 | 54
Eyes
  Grade 0 | 110 | 52
  Grade 1 | 0 | 2
  Grade 2 | 0 | 0
  Grade 3 | 0 | 0
  Grade 4 | 0 | 0

13. Primary Outcome: Number of Eyes With Bulbar Hyperemia - Slit Lamp Findings
Description: Bulbar Hyperemia on slit lamp grading scale 0-4 (0 None: No hyperemia, 1 Trace: Slight regional hyperemia, 2 Mild: Diffuse hyperemia, 3 Moderate: Marked regional or diffuse hyperemia, 4 Severe: Diffuse episcleral or scleral hyperemia)
Time Frame: Baseline
Measure: Number; unit: Eyes
Units Other Than Participants: Eyes
Arm/Group | Invigor A (Test) | Invigor B (Control)
Number analyzed (Participants) | 56 | 28
Number analyzed (Eyes) | 112 | 56
Eyes
  Grade 0 | 88 | 50
  Grade 1 | 24 | 6
  Grade 2 | 0 | 0
  Grade 3 | 0 | 0
  Grade 4 | 0 | 0

14. Primary Outcome: Number of Eyes With Bulbar Hyperemia - Slit Lamp Findings
Description: as for outcome 13
Time Frame: One Month
Population: Two eyes data was not collected for both test and control lens at the one month visit due to lens discomfort.
Measure: Number; unit: Eyes
Units Other Than Participants: Eyes
Arm/Group | Invigor A (Test) | Invigor B (Control)
Number analyzed (Participants) | 55 | 27
Number analyzed (Eyes) | 110 | 54
Eyes
  Grade 0 | 90 | 46
  Grade 1 | 20 | 8
  Grade 2 | 0 | 0
  Grade 3 | 0 | 0
  Grade 4 | 0 | 0

15. Primary Outcome: Number of Eyes With Palpebral Conjunctival Observations - Slit Lamp Findings
Description: Number of Eyes With Palpebral Conjunctival Observations on slit lamp findings - Present / Absent
Time Frame: Baseline
Measure: Number; unit: Eyes
Units Other Than Participants: Eyes
Arm/Group | Invigor A (Test) | Invigor B (Control)
Number analyzed (Participants) | 56 | 28
Number analyzed (Eyes) | 112 | 56
Eyes
  Present | 36 | 20
  Absent | 76 | 36

16. Primary Outcome: Number of Eyes With Palpebral Conjunctiva - Slit Lamp Findings
Description: Palpebral Conjunctival Observations on slit lamp findings - Present / Absent
Time Frame: One Month
Population: Two eyes data was not collected for both test and control lens at the one month visit due to lens discomfort.
Measure: Number; unit: Eyes
Units Other Than Participants: Eyes
Arm/Group | Invigor A (Test) | Invigor B (Control)
Number analyzed (Participants) | 55 | 27
Number analyzed (Eyes) | 110 | 54
Eyes
  Present | 42 | 12
  Absent | 68 | 42

17. Primary Outcome: Number of Eyes With Other Findings - Conjunctival Infection, Epidemic Keratoconjunctivitis, Corneal Ulcers, Iritis, Lens Adhesions and Recurrent Erosion - Slit Lamp Findings
Description: Clinical entities such as conjunctival infection, epidemic keratoconjunctivitis, corneal ulcers, iritis, lens adhesions and recurrent erosion on Slit lamp grading scale of 0-4 (0 None
  1 Trace, 2 Mild, 3 Moderate, 4 Severe)
Time Frame: Baseline
Measure: Number; unit: Eyes
Units Other Than Participants: Eyes
Arm/Group | Invigor A (Test) | Invigor B (Control)
Number analyzed (Participants) | 56 | 28
Number analyzed (Eyes) | 112 | 56
Eyes
  Grade 0 | 112 | 56
  Garde 1 | 0 | 0
  Grade 2 | 0 | 0
  Grade 3 | 0 | 0
  Grade 4 | 0 | 0

18. Primary Outcome: Number of Eyes With Other Findings - Conjunctival Infection, Epidemic Keratoconjunctivitis, Corneal Ulcers, Iritis, Lens Adhesions and Recurrent Erosion - Slit Lamp Findings
Description: as for outcome 17
Time Frame: One Month
Population: Two eyes data was not collected for both test and control lens at the one month visit due to lens discomfort.
Measure: Number; unit: Eyes
Units Other Than Participants: Eyes
Arm/Group | Invigor A (Test) | Invigor B (Control)
Number analyzed (Participants) | 55 | 27
Number analyzed (Eyes) | 110 | 54
Eyes
  Grade 0 | 106 | 52
  Garde 1 | 4 | 2
  Grade 2 | 0 | 0
  Grade 3 | 0 | 0
  Grade 4 | 0 | 0

19. Secondary Outcome: Number of Eyes With Visual Acuity for an Effective Visual Distance of 20 Feet
Description: Number of Eyes With Visual Acuity was assessed using Snellen VA Chart for an effective visual distance of 20 feet
Time Frame: One Month
Population: Two eyes data was not collected for both test and control lens at the one month visit due to lens discomfort.
Measure: Number; unit: Eyes
Units Other Than Participants: Eyes
Arm/Group | Invigor A (Test) | Invigor B (Control)
Number analyzed (Participants) | 55 | 27
Number analyzed (Eyes) | 110 | 54
Eyes
  20/20 | 92 | 45
  20/15 | 7 | 4
  20/25 | 11 | 5

ADVERSE EVENTS:
Time Frame: From dispense up to one month for each study lenses
Arm/Group | Invigor A (Test) | Invigor B (Control)
All-Cause Mortality (participants affected / at risk) | 0/56 | 0/28
Serious Adverse Events (participants affected / at risk) | 0/56 | 0/28
Other Adverse Events (participants affected / at risk) | 0/56 | 0/28

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-10-03): https://cdn.clinicaltrials.gov/large-docs/84/NCT03722784/Prot_SAP_000.pdf